CLINICAL TRIAL: NCT05155488
Title: Mucopolysaccharidosis Type II in Brazil: A Retrospective Secondary Database Study (Informatics Department of Brazilian Health System - DATASUS)
Brief Title: A Study to Improve the Awareness of Mucopolysaccharidosis Type II in Brazil
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-765-5001; MACS-2021-021601 (Other: Takeda)
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Mucopolysaccharidosis (MPS)
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With MPS II: Retrospective data of participants diagnosed with MPS II will be collected from the database (DATASUS) from January 1st, 2008 to September 30th, 2020 in this observational study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aims of the study are to learn about the percentage of mucopolysaccharidosis type II (MPS II) in adults in Brazil as well as about the diagnosis process. No study medicines will be provided to participants in this study. The data available for participants diagnosed with MPS II in DATASUS (a database of the Informatics Department of Brazilian Health System) will be reviewed. No clinic visits will be required as part of participation in this study.

ELIGIBILITY:
Inclusion Criteria:

All MPS II cases of (International Classification of Diseases, 10th revision [ICD-10] E76.1) at any age reported in DATASUS from January 1st, 2008 to September 30th, 2020 will be included.

Exclusion Criteria:

MPS II cases reported outside this period will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with MPS II cases in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants Diagnosed With MPS II | From January 1, 2008 to September 30, 2020
  Number of participants diagnosed with MPS II will be reported based on the retrospective data of participants collected from the database (DATASUS).
Number of Participants with Comorbidities Associated with MPS II | From January 1, 2008 to September 30, 2020
  Comorbidities will be like respiratory infections, carpal tunnel syndrome and hernia. Number of participants with comorbidities associated with MPSII will be reported based on the retrospective data of participants collected from the database (DATASUS).
Age of MPS II Diagnosis | From January 1, 2008 to September 30, 2020
  Age of MPS II diagnosis will be calculated from the date of birth and date of diagnosis. Retrospective data of participants will be collected from the database (DATASUS).

SECONDARY OUTCOMES:
Number of Health Care Professionals Who Diagnosed MPS II | From January 1, 2008 to September 30, 2020
  Number of health care professionals who diagnosed the MPS II will be reported based on the retrospective data of participants collected from the database (DATASUS).
Number of Health Care Professionals Consulted | From January 1, 2008 to September 30, 2020
  Number of health care professionals consulted before MPS II diagnosis will be reported based on the retrospective data of participants collected from the database (DATASUS).
Time to MPS II Diagnoses | From January 1, 2008 to September 30, 2020
  Time between first Unified Health System (a Brazilian Health System) consultation and MPS II diagnosis will be reported based on the retrospective data of participants collected from the database (DATASUS).
Time Between MPS Diagnosis II and Start of Treatment | From January 1, 2008 to September 30, 2020
  Time between MPS diagnosis II and start of treatment will be reported based on the retrospective data of participants collected from the database (DATASUS).
Number of Treatments Received Before and After MPS II Diagnosis | From January 1, 2008 to September 30, 2020
  Number of treatments received by participant before and after MPS II diagnosis will be reported based on the retrospective data of participants collected from the database (DATASUS).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Distribuidora Ltda, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61b7bf0df571d4002a64b48c